CLINICAL TRIAL: NCT06507787
Title: Evaluation of the Impact of the EDIT-B® Blood Test on the Health Status of Patients Presenting a Major Depressive Episode. Clinical Utility and Medico-Economic Aspects
Acronym: SEM EDIT-B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alcediag (Industry)
Collaborators: BPIfrance (Other); Synlab Holding Deutschland GmbH (Industry); GHU Paris Psychiatrie et Neurosciences (Unknown); CH Erstein (Unknown); AP-HP Corentin-Celton (Unknown); Clinique Villa des Roses (Unknown); Clinique Le clos Montaigne (Unknown); Clinique Médicale de Ville d'Avray (Unknown); EPSM 74 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SEM EDIT-B
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Bipolar Disorder; Major Depressive Disorder
Keywords: Clinical Utility; Bipolar Disorder; Major Depressive Disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With EDIT-B test result (Experimental): The investigator will have the EDIT-B® test result to guide the treatment strategy.
  Interventions: Diagnostic Test: EDIT-B test
- Without EDIT-B test result (Placebo Comparator): The investigator will not have the EDIT-B® test result, but EDIT-B® is still performed on participants in the beginning of the study.
  Interventions: Diagnostic Test: EDIT-B test (without giving result)

INTERVENTIONS:
Diagnostic Test: EDIT-B test — EDIT-B® is the first blood test for the differential diagnosis of bipolar disorder (BD) and major depression. It consists of a biological analysis (including targeted RNA sequencing) followed by a software interpretation thanks to an algorithm developed with AI. The test is CE marked, clinically validated on two independent cohorts and shows an excellent performance with a sensitivity and specificity of more than 80%.
  For performing the test, a blood sample of 2.5 ml will be drawn using PAXgene™ Blood RNA tubes (Becton Dickinson, UK) according to the manufacturer's instructions.
  The objective of EDIT-B® is to reduce the time to diagnosis of BD, which is currently 7 years on average. This will improve the patient pathway, thanks to faster access to appropriate care - whether for unipolar or bipolar patients - with a major medical, social and financial impact.
  Arms: With EDIT-B test result
Diagnostic Test: EDIT-B test (without giving result) — EDIT-B® is the first blood test for the differential diagnosis of bipolar disorder (BD) and major depression. It consists of a biological analysis (including targeted RNA sequencing) followed by a software interpretation thanks to an algorithm developed with AI. The test is CE marked, clinically validated on two independent cohorts and shows an excellent performance with a sensitivity and specificity of more than 80%.
  For performing the test, a blood sample of 2.5 ml will be drawn using PAXgene™ Blood RNA tubes (Becton Dickinson, UK) according to the manufacturer's instructions. THE RESULT OF THE TEST WILL NOT BE GIVEN TO THE PARTICIPANT BEFORE THE END OF THE STUDY.
  The objective of EDIT-B® is to reduce the time to diagnosis of BD, which is currently 7 years on average. This will improve the patient pathway, thanks to faster access to appropriate care - whether for unipolar or bipolar patients - with a major medical, social and financial impact.
  Arms: Without EDIT-B test result

SUMMARY:
Depression is one of the most common mental disorders, affecting nearly 10% of men and 20% of women worldwide. It is associated with a significant increase in mortality, mainly due to suicidal behavior. The Diagnostic and Statistical Manual of Mental Disorders (DSM) defines a Major Depressive Episode (MDE) by a combination of at least five different symptoms, with at least one depressed mood or loss of interest. MDEs can occur in isolation or as part of Major Depressive Disorder (MDD) or bipolar disorder (BD). Bipolar disorders affect 2% of the world's population and are defined by episodes of mania (Type I BD) or hypomania (Type II BD) alternating with episodes of depression and periods of remission.

Depression occurring whether in the context of BD or MDD is defined with the same clinical criteria. However, the pharmacological treatments are different in the two groups. In particular, antidepressants prescribed without a thymoregulator in bipolar patients can lead to a worsening of the episode, favoring suicidal behavior or a manic turn.

The average interval between the onset of BD symptoms and appropriate diagnosis is estimated to be approximately 7 years, which delays appropriate management and treatment and increases the risk of suicide.

Biological markers able to differentiate between the different types of depression were lacking before the advent of EDIT-B®; one of the main objectives of this research is to measure the clinical impact of the use of EDIT-B® in the short and medium term on the management of patients with BD and major depression. The health economic aspect will also be considered.

In total, 450 patients in two different groups (EDIT-B® group and control group) will be recruited over a study timeline of 24 months. Study participation is over 6 months with 4 visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a MDE, moderate to severe (DSM V criteria and MADRS score ≥19)
* Age between 18 and 65 years, gender indifferent
* Benefitting from health insurance coverage
* Having signed an informed consent and agreed to follow the study protocol to completion
* Patients for whom there is doubt regarding a bipolar disorder diagnosis, and/or presenting one or more of the following criteria:

  * More than 3 episodes of MDE in personal medical history
  * Psychotic symptoms
  * Family history of bipolar disorder
  * Onset of the first MDE before the age of 25
  * Atypical symptoms or mixed features during depressive episodes
  * Addiction
  * Personal history of suicide attempts
  * Resistance to antidepressants
  * Postpartum depression within 6 months of birth

Exclusion Criteria:

* Depression in the context of schizophrenia or autism spectrum disorder
* Patient with a well-established diagnosis of bipolar disorder
* Patients who is already receiving a mood stabilizer
* Severe somatic diseases that may interfere with the follow-up or associated with treatments at risk of secondary manic decompensation
* Neurodegenerative diseases
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Improvement in depressive symptoms between inclusion and 15-16 weeks visit. | 4 months (from inclusion visit to 15-16 weeks visit)
  Clinically meaningful improvement at week 15-16 in depressive symptoms, defined as a 6-point or greater reduction in MADRS total score from baseline, without a manic switch, defined as an increase in the YMRS total score above 11 from baseline, measured using a composite endpoint.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CH Erstein, Erstein
  - AP-HP Corentin Celton, Issy-les-Moulineaux
  - Etablissement Public de Santé Mentale (EPSM) 74, La Roche-sur-Foron
  - Clinique Villa des Roses, Lyon
  - Clinique Le Clos Montaigne, Montrond-les-Bains
  - GHU Paris Psychiatrie et Neurosciences, Paris
  - Clinique Médicale de Ville d'Avray, Ville-d'Avray